CLINICAL TRIAL: NCT04706702
Title: Implementation of Tele-Exercise for Management of Knee Osteoarthritis in Older Rural Primary Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kushang Patel, Research Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012144
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-EF (Experimental): Tele-EnhanceFitness
  Interventions: Behavioral: Tele-EnhanceFitness

INTERVENTIONS:
Behavioral: Tele-EnhanceFitness — Livestream, instructor-led tele-exercise classes, involving balance, endurance, and strength training

SUMMARY:
Knee osteoarthritis (OA) is highly prevalent and a leading cause of pain that limits physical functioning in older adults. Clinical practice guidelines recommend physical exercise for managing symptoms of knee OA. As a result, several evidence-based exercise programs have been implemented in community centers. However, access to these programs is severely limited in rural settings. Considering that rural communities have a higher disease burden and higher proportion of older adults than non-rural areas, there is a critical need to (1) adapt evidence-based exercise programs for remote delivery to increase access for rural older adults and (2) develop pathways to implement exercise programs in rural health care systems that consistently reach and engage patients with knee OA. Accordingly, we aim to engage rural primary care practices (including medical directors, clinicians, and staff) to develop a clinical pathway that refers patients to an evidence-based exercise program, called Enhance Fitness® (EF), which we have adapted for remote delivery (tele-EF). Enhance Fitness is a group exercise program that is recommended by the CDC for OA management. It is available in over 800 sites nationally and is covered by Medicare Advantage plans, but it is generally not available in rural communities. In addition, we will assess the feasibility and acceptability of implementing the clinical pathway that identifies physically inactive older patients with knee OA, facilitates exercise prescription, and streamlines referral to tele-EF in a rural primary care clinic over a 5-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Community-dwelling
* English-speaking
* Physician diagnosed knee osteoarthritis
* Physically inactive as determined by the 2-item Physical Activity Vital Sign questionnaire

Exclusion Criteria:

* Cognitive impairment determined by a Mini Montreal Cognitive Assessment score of <11
* Significant, non-corrected visual or hearing impairment
* Plans to move out of the area in the next 6 months
* Cancer requiring treatment (except for non-melanoma skin cancer) in the past 6 months
* Heart attack in the past 6 months
* Stroke in the past 6 months
* Hip fracture in the past 6 months
* Hip/knee replacement in the past 6 months
* Spinal surgery in the past 6 months
* Heart surgery in the past 6 months
* Deep vein thrombosis in the past 6 months
* Pulmonary embolus in the past 6 months
* Hospitalization within the last month
* ≥3 falls within the past month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-02-18 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Active minutes per day | Change from Baseline Active Minutes at 12 weeks
  Average number of minutes spent in moderate to vigorous physical activity as measured by the activPAL accelerometer

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function 8-item Short Form | Change from Baseline PROMIS Physical Function score at 12 weeks
  Patient-reported physical functioning
Knee injury and Osteoarthritis Outcome Score (KOOS) Physical Function Subscale | Change from Baseline KOOS Physical Function Subscale score at 12 weeks
  Patient-reported knee pain-related interference with physical functioning

CONTACTS AND LOCATIONS:
Overall Officials: Kushang V Patel, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators recognize that data sharing leads to the promotion of science. We intend to publish the results of the proposed study and will make data available to investigators upon request (following publication). The final dataset will include demographic, clinical, and behavioral data on 15 older adults followed over a 3-month period. Even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that the possibility of deductive disclosure of subjects with unusual characteristics remains. For these reasons, we propose to make the data and associated documentation available to users under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.